CLINICAL TRIAL: NCT03857620
Title: Improving Surgical Care and Outcomes in Older Cancer Patients Through Implementation of an Efficient Pre-Surgical Toolkit (OPTI-Surg)
Brief Title: Use of a Pre-Surgical Toolkit in Improving Surgical Care and Outcomes in Older Participants With Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: A231601CD; NCI-2018-01512 (Registry Identifier: NCI Clinical Trial Reporting Program); UG1CA189823 (NIH)
Record Dates: First submitted 2019-02-26; First posted 2019-02-28 (Actual); Results first posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-01

CONDITIONS: Malignant Neoplasm; Surgical Procedure, Unspecified; Health Care Provider; Carcinoma
MeSH Terms: conditions — Neoplasms; Carcinoma | interventions — Practice Guidelines as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm I (usual care) (Active Comparator): Healthcare providers/institutions perform usual care.
  Interventions: Other: Best Practice; Other: Questionnaire Administration
- Arm II (OPTI-Surg training and materials) (Experimental): Healthcare providers/institutions receive OPTI-Surg training and informational materials.
  Interventions: Other: Informational Intervention; Other: Questionnaire Administration
- Arm III (OPTI-Surg training and materials, coach) (Experimental): Healthcare providers/institutions receive OPTI-Surg training and informational materials and meet with a coach.
  Interventions: Other: Questionnaire Administration; Other: Informational Intervention with Coaching

INTERVENTIONS:
Other: Best Practice — Receive usual care
  Arms: Arm I (usual care)
Other: Informational Intervention — Receive OPTI-Surg program materials
  Arms: Arm II (OPTI-Surg training and materials)
Other: Questionnaire Administration — Ancillary studies
Other: Informational Intervention with Coaching — Receive OPTI-Surg program materials plus individual coaching
  Arms: Arm III (OPTI-Surg training and materials, coach)

SUMMARY:
This trial studies how well the use of a pre-surgical toolkit (OPTI-Surg) works in improving surgical care and outcomes in older participants with cancer. In many elderly patients, surgery can greatly affect physical condition and the ability to return to pre-surgery levels of physical functioning. Providing pre-surgical recommendations may help improve participants' recovery rate and functioning after surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare 8-week postoperative function among elderly patients between sites randomized to implement the OPTI-Surg toolkit with or without a coach versus sites randomized to usual care.

SECONDARY OBJECTIVES:

I. To compare postoperative morbidity between sites randomized to implement the OPTI-Surg toolkit with or without a coach versus sites randomized to usual care.

II. To compare the penetration of the OPTI-Surg toolkit between sites randomized to implement the OPTI-Surg toolkit with a coach versus sites randomized to implement the OPTI-Surg toolkit without a coach.

Trial Design:

OUTLINE: Healthcare providers/institutions are randomized to 1 of 3 arms. Patients/participants receive the intervention based on which arm their healthcare provider is in.

ARM I: Healthcare providers/institutions perform usual care.

ARM II: Healthcare providers/institutions receive OPTI-Surg training and informational materials.

ARM III: Healthcare providers/institutions receive OPTI-Surg training and informational materials and meet with a coach.

After conclusion of study, participants are followed up at 8 and 12 weeks post surgery, and healthcare providers/institutions are followed up 6-9 months after the last patient is registered.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have known or suspected cancer diagnosis and have one of the following cancer-directed operations planned:

  * Gastrectomy
  * Colectomy
  * Proctectomy
  * Esophagectomy
  * Pancreatectomy
  * Hepatectomy
  * Total cystectomy
  * Partial or total nephrectomy
  * Lung lobectomy/pneumonectomy
* Patients with known metastatic disease with a plan for curative intent resection are eligible (e.g. curative liver resection for metastatic colorectal cancer).
* Patients with double primaries undergoing planned curative operation for both are eligible (e.g. synchronous colon cancers undergoing colectomy to treat both).
* Patients must be able to speak and complete questionnaires in English.

Exclusion Criteria:

* Patients undergoing emergent surgery are not eligible.
* Patients under active treatment such as chemotherapy, targeted therapy, immunotherapy, radiation treatment, etc. for second primary, are not eligible.
* Patients with second primary are not eligible.
* Patients with known metastatic disease who are undergoing palliative resection are not eligible.
* Patients with psychiatric illness or other mental impairment that would preclude their ability to give informed consent or to participate in the prehabilitation program are not eligible.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 325 (Actual)
Dates: Start 2019-07-24 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2025-10 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: George J. Chang, MD, MS, Study Chair — M.D. Anderson Cancer Center
Locations (44):
- United States (44):
  - Helen F Graham Cancer Center, Newark, Delaware
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Augusta University Medical Center, Augusta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Queen's Medical Center, Honolulu, Hawaii
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - LSU Healthcare Network / Metairie Multi-Specialty Clinic, Metairie, Louisiana
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Fairview Southdale Hospital, Edina, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Baptist Memorial Hospital and Cancer Center-Desoto, Southhaven, Mississippi
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Morristown Medical Center, Morristown, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Novant Health Forsyth Medical Center, Winston-Salem, North Carolina
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Miami Valley Hospital South, Centerville, Ohio
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - VCU Massey Cancer Center at Stony Point, Richmond, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Ascension Southeast Wisconsin Hospital - Elmbrook Campus, Brookfield, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Ascension Southeast Wisconsin Hospital - Franklin, Franklin, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin

REFERENCES:
- [Derived] Zahrieh D, Croghan IT, Inselman JW, Mandrekar SJ. Guidelines for Data and Safety Monitoring in Pragmatic Randomized Clinical Trials Using Case Studies. Mayo Clin Proc. 2023 Nov;98(11):1712-1726. doi: 10.1016/j.mayocp.2023.02.019. PMID 37923529

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Three-hundred and twenty-five participants (94 Arm I, 114 Arm II, 117 Arm III) were enrolled between April 2019 to September 2022 from 29 sites (10 Arm I, 9 Arm II, 10 Arm III). Recruitment was temporarily paused from March 25, 2020 to June 15, 2020 due to the COVID-19 pandemic. Data as of 3/15/2024 that was summarized for manuscript submission, is reported here.
Pre-assignment Details: This was a cluster-randomized trial at the practice level. Thirty sites with practice types of major abdominal (18 sites), thoracic (6 sites) or urologic (6 sites) were randomized initially in a 1:1:1 fashion to each arm. A total of 9 sites withdrew prior to accruing a patient due to inability to meet accrual expectations/had issues with resource allocation. Eight additional sites were randomized. A total of 29 sites remained with the study participation and accrued at least 1 patient.
Units Other Than Participants: Sites
Period: Overall Study
Arm/Group | Arm I (Usual Care) | Arm II (OPTI-Surg Training and Materials) | Arm III (OPTI-Surg Training and Materials, Coach)
Started | 94; 13 Sites | 114; 14 Sites | 117; 11 Sites
Completed | 68; 10 Sites | 83; 9 Sites | 92; 10 Sites
Not Completed | 26; 3 Sites | 31; 5 Sites | 25; 1 Sites
Not completed — Death | 4 | 5 | 7
Not completed — Lost to Follow-up | 2 | 5 | 3
Not completed — Disease progression or relapse after study registration | 1 | 5 | 1
Not completed — Ineligible | 5 | 0 | 2
Not completed — No malignancy | 1 | 0 | 1
Not completed — Patient withdrawal/refusal prior to surgery | 2 | 0 | 0
Not completed — Patient withdrawal/refusal after surgery performed | 4 | 7 | 2
Not completed — Surgery not performed due to worsening performance status/medical ineligibility | 4 | 4 | 3
Not completed — Surgery not performed, patient decision | 0 | 3 | 1
Not completed — Surgery not performed, other reason | 3 | 1 | 4
Not completed — Worsening performance status after surgery performed | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Usual Care) | Arm II (OPTI-Surg Training and Materials) | Arm III (OPTI-Surg Training and Materials, Coach) | Total
Number analyzed (Participants) | 94 | 114 | 117 | 325
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.5 (4.83) | 75.6 (4.73) | 76.7 (5.12) | 76.3 (4.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 50 | 55 | 148
  Male | 51 | 64 | 62 | 177
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 4 | 0 | 8 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 4 | 4
  Black or African American | 7 | 13 | 12 | 32
  White | 80 | 97 | 86 | 263
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3 | 4 | 6 | 13
Region of Enrollment [Number; unit: participants]
  United States | 94 | 114 | 117 | 325
Baseline Weight [Mean (Standard Deviation); unit: kg] | 77.1 (13.47) | 81 (18.68) | 82.4 (20.38) | 80.4 (18.06)

OUTCOME MEASURES:

1. Primary Outcome: Physical Function 8 Weeks Post-surgery as Measured by the Caloric Expenditure Scale Per Community Healthy Activities Model Program for Seniors (CHAMPS) Questionnaire
Description: The CHAMPS questionnaire includes 41 questions that measures frequency and duration of activities. The primary endpoint is the estimated Caloric Expenditure Per Week measure from the CHAMPS, which is calculated by weighting the duration variable of the 28 exercise-related activities using the corresponding metabolic equivalents (METs) value, then multiplying by 60 to convert METs/minute to METs/hour, then multiplying by participant weight in kg/200 to calculate the caloric expenditure/week score, and then summing the individual item caloric expenditure scores across all 28 items. This scale score was transformed into the unit of kcal. The minimum possible value of the scale is 0 and there is not a defined maximum possible value. Higher scores equate to more kilocalories burned per week, which is a better outcome in the context of this trial.
Time Frame: 8 weeks post surgery
Population: All eligible participants who undergo major cancer surgery, consent to complete CHAMPS questionnaires, have a baseline CHAMPS score and have a CHAMPS score at 8 weeks post-surgery +/- 2 weeks.
Measure: Mean (Standard Deviation); unit: kcal
Arm/Group | Arm I (Usual Care) | Arm II (OPTI-Surg Training and Materials) | Arm III (OPTI-Surg Training and Materials, Coach)
Number analyzed (Participants) | 64 | 68 | 67
kcal
  Baseline | 2.5 (2.53) | 2.3 (2.45) | 3.0 (2.96)
  8 weeks post-surgery | 2.2 (1.94) | 2.2 (2.26) | 1.9 (1.76)
Statistical Analysis 1: Comparison: Arm I (Usual Care) vs Arm II (OPTI-Surg Training and Materials) vs Arm III (OPTI-Surg Training and Materials, Coach); Combined Arm II (OPTI-Surg) & Arm III (OPTI-Surg plus Coach) vs. Arm I (Usual Care); Test type: Superiority; p = 0.53, Mixed Models Analysis; Generalized linear mixed effects model (w/ Gaussian link) w/ random practice effect to account for clustering by site & bsl CHAMPS score as covariate; Mean Difference (Final Values) = -0.20, 95% CI 2-sided [-0.85 to 0.45]
Statistical Analysis 2: Comparison: Arm I (Usual Care) vs Arm II (OPTI-Surg Training and Materials); Test type: Superiority; p = 0.84, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.07, 95% CI 2-sided [-0.67 to 0.81]
Statistical Analysis 3: Comparison: Arm I (Usual Care) vs Arm III (OPTI-Surg Training and Materials, Coach); Test type: Superiority; p = 0.19, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.48, 95% CI 2-sided [-1.21 to 0.26]
Statistical Analysis 4: Comparison: Arm II (OPTI-Surg Training and Materials) vs Arm III (OPTI-Surg Training and Materials, Coach); Test type: Superiority; p = 0.14, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.55, 95% CI 2-sided [-0.19 to 1.29]

2. Secondary Outcome: Percentage of Participants With Postoperative Complications (Clavien-Dindo Grades I-V)
Description: Postoperative complications were assessed at 12 weeks following surgery using the Clavien-Dindo classification:
  Grade I: Any deviation from the normal postoperative course w/out the need for pharmacological treatment or surgical, endoscopic, and radiological interventions Grade II: Requiring pharmacological treatment w/ drug other than such allowed for Grade I complications Grade III: Requiring surgical, endoscopic or radiological intervention Grade IIIa: Intervention not under general anesthesia Grade IIIb: Intervention under general anesthesia Grave IV: Life-threatening complication Grade IVa: Single organ dysfunction Grade IVb: Multiorgan dysfunction Grave V: Death A generalized linear mixed model (with logit link function) with random practice effect to account for clustering within practice will be used to compare postoperative complications within 12 weeks of surgery between the combined OPTI-Surg no-coach & coach arms vs usual care followed by pairwise comparisons
Time Frame: 12 weeks
Population: All eligible participants who undergo major cancer surgery (no documentation of postoperative complications will be considered as not having any postoperative complications).
Measure: Number; unit: percentage of participants
Arm/Group | Arm I (Usual Care) | Arm II (OPTI-Surg Training and Materials) | Arm III (OPTI-Surg Training and Materials, Coach)
Number analyzed (Participants) | 78 | 96 | 105
percentage of participants | 25.6 | 44.8 | 26.7
Statistical Analysis 1: Comparison: Arm I (Usual Care) vs Arm II (OPTI-Surg Training and Materials) vs Arm III (OPTI-Surg Training and Materials, Coach); Combined Arm II (OPTI-Surg) & Arm III (OPTI-Surg plus Coach) vs. Arm I (Usual Care); Test type: Superiority; p = 0.50, Mixed Models Analysis; Generalized linear mixed effects model (with logit link function) with a random practice effect to account for clustering within practice; Odds Ratio (OR) = 0.70, 95% CI 2-sided [0.23 to 2.09]
Statistical Analysis 2: Comparison: Arm I (Usual Care) vs Arm II (OPTI-Surg Training and Materials); Test type: Superiority; p = 0.21, Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 0.46, 95% CI 2-sided [0.13 to 1.62]
Statistical Analysis 3: Comparison: Arm I (Usual Care) vs Arm III (OPTI-Surg Training and Materials, Coach); Test type: Superiority; p = 0.96, Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 1.03, 95% CI 2-sided [0.30 to 3.54]
Statistical Analysis 4: Comparison: Arm II (OPTI-Surg Training and Materials) vs Arm III (OPTI-Surg Training and Materials, Coach); Test type: Superiority; p = 0.19, Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 0.45, 95% CI 2-sided [0.13 to 1.54]

3. Secondary Outcome: Compliance Rate With Administration of Edmonton Frail Scale (EFS)
Description: EFS is a validated measure of frailty that identifies distinct frailty domains that are potential targets for additional pre-operative optimization. For frailty domains that score 1 or 2 points, optimization referrals will be recommended. Clinic or research staff at sites randomized to OPTI-Surg intervention arms will screen and identify eligible patients for administration of the EFS and provide printed surgery preparation materials. A generalized linear mixed model (with logit link function) with a random practice effect to account for clustering within practice will be used to compare compliance rate for screening between the no-coach and coach arms.
Time Frame: Day of surgical consult
Population: All eligible participants from Arm II (OPTI-Surg) and Arm III (OPTI-Surg plus Coach) who undergo major cancer surgery who are evaluable for postoperative complications outcome. Notes: Generalized linear mixed model analysis not performed.
Measure: Number; unit: percentage of participants
Arm/Group | Arm II (OPTI-Surg Training and Materials) | Arm III (OPTI-Surg Training and Materials, Coach)
Number analyzed (Participants) | 96 | 105
percentage of participants | 99 | 100

ADVERSE EVENTS:
Time Frame: Duration of the study, up to 1 year
Description: The exclusion to CTEP-AERS Expedited Reporting Requirements was outlined in the study Protocol Section 9.3.3. The adverse events were assessed only between initial surgical consultation (baseline) and on the day of surgery and additional reporting per Section 9.3.3. The study intervention refers to the administration of the OPTI-Surg toolkit (Edmonton Frail Scale and the follow-up recommendations) and not the surgery itself, which is why this trial doesn't have a typical collection of AEs.
Arm/Group | Arm I (Usual Care) | Arm II (OPTI-Surg Training and Materials) | Arm III (OPTI-Surg Training and Materials, Coach)
All-Cause Mortality (participants affected / at risk) | 4/94 | 5/114 | 7/117
Serious Adverse Events (participants affected / at risk) | 0/94 | 3/114 | 3/117
Other Adverse Events (participants affected / at risk) | 5/94 | 16/114 | 13/117
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Usual Care) (N=94) | Arm II (OPTI-Surg Training and Materials) (N=114) | Arm III (OPTI-Surg Training and Materials, Coach) (N=117)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Heart failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Intestinal stoma leak (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Death NOS (General disorders) | 0 (0) | 2 (2) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Usual Care) (N=94) | Arm II (OPTI-Surg Training and Materials) (N=114) | Arm III (OPTI-Surg Training and Materials, Coach) (N=117)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 13 (13) | 2 (2)
Lymphocyte count decreased (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Arterial fibrilation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac disorders - Other, specify (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Obstruction gastric (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pancreatic fistula (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Fever (General disorders) | 0 (0) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 1 (1)
Gen disord and admin site conds-Oth spec (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
Esophageal anastomotic leak (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Cholesterol high (Investigations) | 0 (0) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 9 (9) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 4 (4) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Renal and urinary disorders - Oth spec (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Surgical and medical proced - Oth spec (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 1 (1) | 4 (4)
Hypotension (Vascular disorders) | 1 (1) | 2 (2) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-09-16): https://cdn.clinicaltrials.gov/large-docs/20/NCT03857620/Prot_SAP_ICF_000.pdf